CLINICAL TRIAL: NCT04916275
Title: Stress Post Traumatique, Signes de dépression et Syndrome d'épuisement Professionnel Chez le Personnel Des EHPAD en Occitanie Pendant la pandémie COVID-19 : étude Prospective
Brief Title: Post-traumatic Stress, Signs of Depression and Burnout Syndrome Among Nursing Home Staff in Occitanie During the COVID-19 Pandemic
Acronym: PSY-COEHPAD-OC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2020/COVID/JYL IC-04; 2020-A03541-38 (Other: ANSM)
Record Dates: First submitted 2021-06-04; First posted 2021-06-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Post Traumatic Stress Disorder; Anxiety; Depressive Disorder; Substance Use Disorders
MeSH Terms: conditions — COVID-19; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depressive Disorder; Substance-Related Disorders | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Staff working in a nursing home in Occitanie
  Interventions: Other: Cognitive tests

INTERVENTIONS:
Other: Cognitive tests — Optional tests: Corsi block-tapping task, Stroop test and Iowa gambling task

SUMMARY:
Nursing home staff face multiple stresses during the Covid-19 pandemic including personal risk of infection, risk of transmission of the virus to residents and relatives, and risk of witnessing end-of-life scenarios under difficult contexts (absence of families). The hypothesis of this study is that the Covid-19 period is associated with an incidence of more than 30% of post-traumatic stress in nursing home staff.

ELIGIBILITY:
Inclusion Criteria:

* Professional working in a nursing home in Occitanie
* Professional agreeing to participate
* Professional in a nursing home for at least 3 months
* Professional able to read French
* Profession with an internet connection

Exclusion Criteria:

* The subject is in a period of exclusion determined by a previous study
* The subject refuses to participate
* The subject has already been included into the study
* It is impossible to give the subject informed information
* The subject is under safeguard of justice or state guardianship
* The subject is unable to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Professionasl working in a nursing home in Occitanie
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
To assess the prevalence of post-traumatic stress disorder (PTSD) in the context of the COVID-19 health crisis | Day 0
  Posttraumatic Stress Disorder Checklist Scale (PCL-5) scale, where the recommended cut-off threshold for screening is 44

SECONDARY OUTCOMES:
Prevalence of depression in the context of the COVID-19 health crisis | Day 0
  Hospital Anxiety and Depression Scale (HADS) scale, using a cut-off above 7
Prevalence of burn out in the context of the COVID-19 health crisis | Day 0
  Masslach Burn out Inventory (MBI) questionnaire where high scores for the professional burnout and depersonalization sections and a low score for the personal accomplishments section will signal burn out

OTHER OUTCOMES:
Optional assessment of work memory abnormalities associated with symptoms of post-traumatic stress disorder, anxiety and depression | Day 0
  Corsi block-tapping task - score ranging from 0(good memory) -18(bad memory)
Optional assessment of cognitive flexibility abnormalities associated with symptoms of post-traumatic stress disorder, anxiety and depression | Day 0
  Corsi block-tapping task - score ranging from 0(good memory) -18(bad memory)
Optional assessment of decision-making abnormalities associated with symptoms of post-traumatic stress disorder, anxiety and depression | Day 0
  Iowa Gambling Task - score ranes from -14 to +40

CONTACTS AND LOCATIONS:
Overall Officials: Ismaël Conejero, Principal Investigator — CHU de Nimes
Locations (3):
- France (3):
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Hôpital Universitaire Carémeau, Nîmes
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Result] Conejero I, Petrier M, Fabbro Peray P, Voisin C, Courtet P, Potier H, Elotmani L, Lafont B, Lefrant JY, Lopez Castroman J, Arbus C, Blain H. Post-traumatic stress disorder, anxiety, depression and burnout in nursing home staff in South France during the COVID-19 pandemic. Transl Psychiatry. 2023 Jun 15;13(1):205. doi: 10.1038/s41398-023-02488-1. PMID 37322006